CLINICAL TRIAL: NCT02418923
Title: HemoSonics-UVA Spinal Surgery Clinical Study Protocol
Brief Title: HemoSonics-UVA Spinal Surgery
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: HemoSonics LLC (Industry)
Responsible Party: Principal Investigator, Bhiken I. Naik, MD, UVA Anesthesiology Faculty, University of Virginia
Other Study IDs: 17942
Record Dates: First submitted 2015-04-13; First posted 2015-04-17 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Deformity of Spine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Procedure: Blood specimen collection — Blood specimen collection

SUMMARY:
This study compares the results of current standard coagulation measurement devices to the Quantra System, a new device, using small amount of extra blood obtained during routine blood draws in neurosurgery patients.

DETAILED DESCRIPTION:
HemoSonics is developing a novel POC diagnostic device, the Quantra System, to perform whole blood coagulation analysis and which is suitable for use in surgical and intensive care settings. The Quantra System employs a patented technology named sonorheometry, which was invented at the University of Virginia.

Sonorheometry uses ultrasound pulses to characterize the dynamic changes in viscoelastic properties of a blood sample during coagulation and clot lysis. The initial assay performed on the Quantra System will be the surgical assay for monitoring hemostasis during major surgical procedures in adult patients.

A clinical study will be conducted to evaluate the analytical performance as well as compared to existing coagulation monitoring technology

ELIGIBILITY:
Inclusion Criteria:

* • Subject is scheduled for major deformity correction spine surgery

  * Subject is older than 18 years
  * Subject is willing to participate and he/she has signed a consent form

Exclusion Criteria:

* • Subject is unable to provide written informed consent

  * Subject is incarcerated at the time of the study
  * Subject is affected by any condition that, in the opinion of the surgical team, may pose additional risks
  * Subjects with renal disease (defined as serum creatinine greater than 1.5 mg/dl)
  * Subjects with history of active liver disease
  * Subjects affected by Factor V Leiden mutation
  * Subjects affected by von Willebrand disease
  * Subjects with an history of thrombotic disease (more than one DVT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited at the University of Virginia Medical Center. The subject population will be representative of the local racial and ethnic population.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
assay inter-instrument variability | 1 day
  Demonstrate assay inter-instrument variability below 15%
Establish normal ranges | 1 day
  Establish normal ranges

CONTACTS AND LOCATIONS:
Overall Officials: Bhiken Naik, MD, Principal Investigator — UVA Anethesiology Faculty
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No